CLINICAL TRIAL: NCT01585480
Title: Preventing Obesity in the Worksite: A Multi-Message, Multi-"Step" Approach
Acronym: Go!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Healthy Foods Healthy Lives (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1002S78225
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Obesity
Keywords: Obesity; Weight Gain Prevention; Workplace; Intervention; Diet; Exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- weight gain prevention intervention (Experimental)
  Interventions: Behavioral: Weight Gain Prevention Intervention
- No treatment comparison group (No Intervention)

INTERVENTIONS:
Behavioral: Weight Gain Prevention Intervention — 1. Behavioral Approaches
     1. Distribution of pedometers
     2. Traffic light labeling in worksite cafeteria and vending machines
  2. Informational & Persuasive Messages
     1. Stair use prompts
     2. Posters, pamphlets, table toppers
     3. Website
  3. Social Approaches
     a. Identification and training of influential employees (Peer Helpers) to shape healthy norms
  4. Environmental Changes
     1. Traffic light labeling
     2. 1/2 portions at 1/2 price
     3. Walking routes
     4. Introduction of healthier foods
     5. Rearrangement of foods in the cafeteria
     6. Adjusting serving spoon size
  Arms: weight gain prevention intervention

SUMMARY:
The purpose of this research study is to develop, implement, and evaluate a multi-component obesity prevention program in a workplace setting. A quasi-experimental design will be utilized, with hospital employees receiving the intervention and clinic employees serving as the comparison group. It is hypothesized that the intervention group will see greater changes in healthier eating, increased participation in physical activity, and reduced risk for obesity (weight, BMI, waist circumference).

DETAILED DESCRIPTION:
Over one-third of Americans are now considered obese. Efforts to prevent obesity involve changing the individual behaviors that contribute to obesity, mainly healthful eating and physical activity, as well as the social and physical context in which those behaviors take place. Due to their existing networks and available resources, worksites are a logical place to help individuals make healthy choices through health promotion efforts. The purpose of this project is to partner with a community hospital to plan, implement, and evaluate a multi-component obesity prevention program in their workplace. The prevention program will target individual and interpersonal determinants of eating behavior and physical activity, as well as the context in which these behaviors take place. This intervention will include four integrated components: (1) nutrition labeling (using stoplights, calories, and step equivalents) in the worksite cafeteria, and modifying the cafeteria environment, (2) distributing pedometers to employees, (3) persuasive media messaging, and (4) the use of "influentials" to address social norms around eating and physical activity behaviors. A quasi-experimental design will examine the effectiveness of this multi-component worksite obesity prevention program.

ELIGIBILITY:
Inclusion Criteria:

* Employee at one of the hospital/clinic locations participating in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline, 6 months, 12 months
Change in Waist Circumference | Baseline, 6 months,12 months

SECONDARY OUTCOMES:
Eating Behaviors | Baseline, 6 months, 12 months
  Eating behaviors will be assessed by the Multifactor Screener (self-report questionnaire) and food purchase data (objective).
Physical Activity | Baseline, 6 months, 12 months
  Physical Activity will be assessed by multiple self-report measures (Godin Leisure Time Exercise Questionnaire, International Physical Activity Questionnaire, and questions about stair use and steps). Stair use will also be assessed by naturalistic observation.

CONTACTS AND LOCATIONS:
Overall Officials: Lara J LaCaille, PhD, Principal Investigator — University of Minnesota; Jennifer F Schultz, PhD, Principal Investigator — University of Minnesota
Locations (1):
- St. Luke's Hospital and Clinics, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LaCaille LJ, Schultz JF, Goei R, LaCaille RA, Dauner KN, de Souza R, Nowak AV, Regal R. Go!: results from a quasi-experimental obesity prevention trial with hospital employees. BMC Public Health. 2016 Feb 19;16:171. doi: 10.1186/s12889-016-2828-0. PMID 26893128